CLINICAL TRIAL: NCT04741685
Title: Clinical Efectivity of Two Different Sensor-augmented Pumps With Low Predictive Suspension Function
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Principal Investigator, Jesús Moreno Fernández, Principal investigator, Castilla-La Mancha Health Service
Other Study IDs: C-380
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- SAP with LGS: Type 1 diabetes adults patients treated with sensor-augmented insulin pump with low glucose predictive suspension function
  Interventions: Device: TTSX2; Device: MM640G

INTERVENTIONS:
Device: TTSX2 — Treatment with Tandem T Slim X2 with Basal IQ
Device: MM640G — Treatment with Medtronic Minimed 640G with Smartguard

SUMMARY:
Observational cross-sectional multicenter study about effectiveness of two different sensor augmented-pumps with low glucose predictive function in Type 1 Diabetes Mellitus (T1DM) adult patients in routine clinical practice.

DETAILED DESCRIPTION:
Cross-sectional multicenter analysis about clinical effectiveness of two different sensor-augmented pumps, Tandem T Slim X2 with Basal IQ (TTSX2) and Medtronic Minimed 640G with Smartguard (MM640G) in adult patients with type 1 Diabetes mellitus.

All clinical variables are gathered from three EMR softwares and two sensor-augmented pumps sotwares.

Data analysis is conducted using SPSS (Chicago, IL) statistics software. Results are presented as mean ± SD values or percentages. A Kruskal-Wallis or a Friedman test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A "P" value < 0.05 was considered statistically significant.

The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee. All participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Treated with TTSX2 or MM640.

Exclusion Criteria:

* Other kind of diabetes.
* Serious mental disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes adult patients treated with sensor-augmented pump (TTSX2 or MM640G)
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
TIR | during the procedure
  time in range (TIR, 70-180 mg/dL, 3.9-10 mmol/L) of the interstitial glucose

SECONDARY OUTCOMES:
TBR | during the procedure
  time below range (TBR, <70 mg/dL, <3.9 mmol/L) of the interstitial glucose
TAR | during the procedure
  time above range (TIR, 70-180 mg/dL, 3.9-10 mmol/L) of the interstitial glucose
HbA1C | during the procedure
  Glycate haemoglobina A1C
GMI | during the procedure
  Glucose management index
MAGE | during the procedure
  Mean amplitude glucose excursions
%CV | 14 days
  Coefficient of variation percentage of the intersticial glucose
DQOL | during the procedure
  Diabetes quality of life (EsDQOL questionnary score), 43 questions, each question with a score from 1 to 5, worse score is five points.
Hypoglycemia perception 1 | during the procedure
  Hypoglycemia unawareness (Clarke questionnary score), 8 questions, each one score "R" or "not R", more "R" means worse score.
Hypoglycemia perception 2 | during the procedure
  Hypoglycemia unawareness (Gold questionnary scores), single question, score from 0 to 5, worse score is five points.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Nuestra Señora de la Candelaria University Hospital, Santa Cruz de Tenerife, Santa Cruz De Tenerife
  - Badajoz University Hospital, Badajoz
  - Obispo Rafael Torija, St., Ciudad Real

IPD SHARING:
Plan to Share IPD: Undecided
All clinical data if requested.

REFERENCES:
- [Derived] Moreno-Fernandez J, Beato-Vibora P, Olvera P, Garcia-Seco JA, Gallego-Gamero F, Herrera MT, Munoz-Rodriguez JR. Real-world outcomes of two different sensor-augmented insulin pumps with predictive low glucose suspend function in type 1 diabetes patients. Diabetes Res Clin Pract. 2021 Nov;181:109093. doi: 10.1016/j.diabres.2021.109093. Epub 2021 Oct 13. PMID 34653567